CLINICAL TRIAL: NCT04817462
Title: Liver Biopsy In Haemophilia Gene Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18/0130
Record Dates: First submitted 2021-02-23; First posted 2021-03-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hemophilia B, Severe; Hemophilia A, Severe
MeSH Terms: conditions — Hemophilia B; Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Biopsy (Experimental): All patients undergo a liver biopsy only
  Interventions: Procedure: Liver biopsy

INTERVENTIONS:
Procedure: Liver biopsy — The study population is patients with either haemophilia A or B who have previously been administered gene therapy treatment in one of three specific gene therapy clinical trials. In this study they will have a liver biopsy performed to take up to 3 samples for laboratory analysis.

SUMMARY:
To perform a liver biopsy in haemophilia A and B patients with endogenous FVIII:C/FIX:C expression at >1% any time after gene transfer following AAV mediated gene transfer. This is to obtain tissue for analysis, to understand if FIX/FVIII transgenic protein expression is mediated by AAV proviral DNA that is integrated into the host cell DNA or if stable expression in humans is mediated by episomal maintained AAV genome.

DETAILED DESCRIPTION:
To better understand the consequences of AAV gene transfer patients will be recruited to undergo a liver biopsy. Patients will have endogenous FVIII:C/FIX:C expression at >1% any time after gene transfer following AAV mediated gene transfer. Analysis of biopsy samples will:

* Provide a clearer insight into the AAV life cycle in human liver
* Define the number of human hepatocytes that are transduced
* Improve understanding at the human hepatocyte level of long-term consequences of AAV mediated transgene expression from the liver that will include (i) changes in the pattern of gene expression in human hepatocytes following AAV mediated gene transfer, (ii) information on the epigenetic signature in the liver following AAV mediated gene transfer and how this changes with time and (iii) the consequences of transgene expression in hepatocytes.

This study will provide new data addressing several unknowns with AAV mediated gene transfer in humans that will better inform on safety and efficacy following AAV gene transfer for patients who have already participated in gene therapy studies as well as those considering this treatment option.

ELIGIBILITY:
Inclusion criteria:

1. Male and aged 18 to 80 years old
2. Patients who were enrolled and treated in one of the following clinical trials at Royal Free Hospital:

   * AGT4HB (EudraCT No 2005-005711-17) - FIX AAV gene therapy trial (Sponsor: St Jude Children's Research Hospital)
   * GO-8 (EudraCT No 2016-000925-38) - FVIII AAV gene therapy trial (Sponsor: UCL)
   * FLT180a-01 (EudraCT: 2017-000852-24) - FIX AAV gene therapy trial ((Sponsor: UCL) [now enrolled in long term follow up study FLT180a-04 (EudraCT No 2017-005080-40) (Sponsor: Freeline Therapeutics Ltd)
3. Patients with endogenous FVIII:C/FIX:C expression at >1% any time after gene transfer, associated with normal prothrombin (PT) and thrombin times (TT) as determined in a coagulation assay.

Exclusion Criteria:

1. Patients with a platelet count measured at <140 x109/L
2. Any condition that, in the opinion of the investigator or Sponsor would prevent the patient from fully complying with the requirements of the study and/or would influence or interfere with evaluation and interpretation of subject safety or efficacy result.
3. Patients with abnormal kidney function (estimated GFR <50ml/min)
4. Patients with a known allergy to iodine-based intravenous contrast agents
5. Patients with a known allergy to local or general anaesthetic
6. Patients with a known reaction to FVIII/FIX concentrate infusions
7. Presence of FVIII or FIX inhibitor (done within 14 weeks of biopsy)
8. Evidence of any bleeding disorder not related to haemophilia A or B
9. Patients unable and unwilling to provide and sign an informed consent.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of AAV integration in hepatocytes using Target Enrichment Sequencing | Biopsy samples will be taken from participants who are between one month and up to 15 years post gene therapy
  The determination of AAV integration sites will be performed for each participant using Target Enrichment Sequencing (TES) analysis of their liver biopsy sample. This will identify DNA sequences flanking the vector genome. The sequencing data will be analyzed to determine
  1. Vector-Vector Concatemers and Vector-Genome Junctions Analysis
  2. Integration Site,read count, genomic position and nearest gene

SECONDARY OUTCOMES:
Histology analysis using hematoxylin and eosin staining and immunohistochemical staining to determine histopathological changes in hepatocytes | Biopsy samples will be taken from participants who are between one month and up to 15 years post gene therapy
  Hematoxylin and eosin staining and immunohistochemical staining will be done on a liver biopsy sample from each participant to provide information about the structure and distribution of cells and any morphological changes within the liver biopsy sample.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Batty, MBBS MRCP, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom